CLINICAL TRIAL: NCT02394444
Title: Impact of a Psychological Post-hospital Intervention Aimed at Facilitating Parents-child Attachment and Preventing the Preterm Infants' Psycho-emotional, Social and Cognitive Disturbances
Brief Title: Impact of an Intervention Program on Parenting Stress After Preterm Birth
Acronym: IDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Ministry of Health, France (Other Government); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 05-094; 2006/0215 (Registry Identifier: DGS); 2005-36 (Registry Identifier: CPP)
Record Dates: First submitted 2015-02-05; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Preterm Birth; Parenting; Mental Health Wellness 1; Parent-Child Relation; Child Development
Keywords: Intervention program; Parenting stress; Parental mental health; Preterm infant's development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Preterm intervention TRT group (Experimental): Parents with premature infants received the intervention called "Triadic parent-infant's Relationship Therapy" (TRT) :
  the psychological intervention included home visits twice month during the first four months and then monthly visits in the neonatal ward until the 18 months corrected age resulting in a total of 22 visits during the whole intervention; TRT gave attention to emotional distress and the promotion of parenting skills and attachment security; The three sessions of intervention targeted objectives specific to each child's development; A basic manual was designed to ensure uniformity of the defined themes during each session
  Interventions: Other: Triadic parent-infant Relationship Therapy (TRT)
- Preterm control group (No Intervention): Parents with premature infants without intervention program TRT (Triadic parent-infant's Relationship Therapy) received routine follow-up medical care with monthly visits to a practitioner for the first six months and then very three months
- Full-term control group (No Intervention): Parents with full-term infants without intervention program TRT

INTERVENTIONS:
Other: Triadic parent-infant Relationship Therapy (TRT) — 22 sessions, including home visits twice per month during the first four months, followed by monthly consultations in the neonatology ward, up to corrected age of 18 months.
  Other Names: TRT
  Arms: Preterm intervention TRT group

SUMMARY:
The aim of this study was to assess the impact of an early psychological intervention, Triadic parent-infant Relationship Therapy (TRT), on parenting stress, parental mental health, and preterm infant development in the motor, cognitive, emotional and behavioral domains at a corrected age of 18 months.

DETAILED DESCRIPTION:
Due to prematurity induced infant-mother separation at birth, sometimes for several weeks, and owing to the concerns it generates, preterm birth exposes the parent-child attachment link to disturbances, especially the mother-child attachment after discharge. Several psychological factors affect infant (distress, dysmaturity ) and parents (psychological pain). These can cause lasting parent-child interactions disruption and jeopardize the attachment process. These early link distortions may hinder the infant's behavioral-emotional and cognitive development. Prematurity psychological consequences may negatively influence biomedical risks. Understanding these premature infants' future development modalities and support involves taking into account intricate organic and psychological factors - which may be combined as well.

Post-hospital psychological intervention with the family, focusing on parental mental health and triadic parent-infant relationship, proves an essential element in these children care, whose birth conditions were painful.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled preterm infant were required to be between 28 and 35 weeks gestational age +6 days
* Enrolled the parents were required to be French speakers, over 18 years old and residing within 50-kilometres radius of hospital

Exclusion Criteria:

* preterm infant without congenital anomalies or any other foreseeable disabilities during the neonatal period
* parents without known psychiatric history

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2006-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in the "Parent-Infant Relationship" assessed by Parenting Stress Index ( PSI-SF) scores : assessing level of stress in parenting | assessments at each time point: at the corrected ages of 3 and 18 months
Change in "Parent-Infant Relationship" assessed by "R" interview scores : assessing level of parental self-esteem | assessments at each time point: at the corrected ages of 3 and 18 months
"Parent-Infant Relationship" assessed by Q-sort attachment scores : assessing the score of the attachment security of the infant at the corrected age of 18 months | assessment at the corrected age of 18 months
  We needed to use a variety of measures because these measures had to be tailored to the child's stage of development. To ensure the relative strength conclusion on the treatment effect, the statistic analyses of test scores each time point were made using bonefferoni correction for multiple comparisons.
  Parenting Stress Index ( PSI-SF), "R" interview and Q-sort attachment were tests based on the infant's age at different assessment periods.

SECONDARY OUTCOMES:
Change in "Parental Mental Health" assessed by Post-Traumatic Stress Disorder (PTSD) scores: assessing level of post-traumatic stress | assessments at each time point: at 44 weeks gestational age and at the corrected age of 18 months
Change in "Parental Mental Health" assessed by Beck Depression Inventory (BDI) scores: assessing level of depression | assessments at each time point: at 44 weeks gestational age and at the corrected ages of 3, 9 and18 months
Change in "Parental Mental Health" assessed by Edinburgh Postnatal Depression Scale (EPDS) scores: assessing level of postpartum depression | assessments at each time point: at 44 weeks gestational age and at the corrected ages of 3, 9 and18 months
  The BDI and the EPDS are both based on the frequency of depressive symptoms The statistic analyses were used to compare the evolution of all of the other scores over time.
  The Post-Traumatic Stress Disorder (PTSD), Beck Depression Inventory (BDI), Edinburgh Postnatal Depression Scale (EPDS) were tests that were resorted to enable us to examine and monitor the preterm birth traumatic impact on parental mental health.
"Infant Development" assessed by the Neonatal Behavioral Assessment Scale (NBAS) scores: assessing the baby's neurobehavioral development | assessments at 44 weeks gestational age
Change in "Infant Development"assessed by the Brunet-Lezine Psychomotor Development Scales: assessing developmental quotient (DQ) | assessments at each time point: at the corrected ages of 3, 9 and 18 months
Change in "Infant Development"assessed by Infant Behavioral Symptom scores:assessing scores behaviors and emotional capabilities | assessments at each time point: at the corrected ages of 9 and 18 months
  The statistic analyses were used to compare the evolution of all of the other scores over time.
  The Neonatal Behavioral Assessment Scale (NBAS),the Brunet-Lezine Psychomotor Development Scale and Infant Behavioral Symptom were tests that were complementary and enable us to assess infant's various facets of socio-emotional, motor and cognitive development at different stage of development.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Guillois, PhD, Principal Investigator — Neonatology Department, Hospital and university center, Caen; Sophie Castel, MD, Principal Investigator — Neonatology Department, Hospital and university center, Caen

REFERENCES:
- [Background] Guillois B, Castel S, Beunard A, Blaizot X, Creveuil C, Proia-Lelouey N. [Effect of early intervention programs on neurobehavioral outcome in premature infants after discharge]. Arch Pediatr. 2012 Sep;19(9):990-7. doi: 10.1016/j.arcped.2012.06.004. Epub 2012 Aug 9. French. PMID 22884746
- [Background] Sizun, J., Guillois, B., Casper, C., Thiriez, G., Kuhn, P. 2014.Soins de développement en période néonatale.De la recherche à la pratique. Springer.
- [Background] This study was submitted at the 52nd Annual Meeting of the European Society for Pediatric Research at Newcastle (october 15-17th 2011)
- [Background] This study was presented in Communication at the 42nd Journées Nationales de Néonatologie in Paris, march 2012.